CLINICAL TRIAL: NCT02157415
Title: Prospective Cohort Study on the Tolerability and Safety of Uro-Tainer® Polihexanide 0.02% in Long-term Indwelling Catheterized Patients.
Brief Title: Prospective Cohort Study on Tolerability & Safety of Uro-Tainer® Polihexanide 0.02%
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After consultation with a medical expert the Notified Body confirmed premature termination of the study.
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPM-G-H-1101; Cl V-1 3-03-010344 (Other: EUDAMED)
Record Dates: First submitted 2014-05-09; First posted 2014-06-06 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Complications; Catheter, Urinary (Indwelling Catheter) (Suprapubic)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Long-term catherized patients (Experimental): Uro-Tainer Polihexanide 0.02% 100ml rinsing solution
  Interventions: Device: Uro-Tainer Polihexanide 0.02%

INTERVENTIONS:
Device: Uro-Tainer Polihexanide 0.02% — Catheters will be rinsed by gravity feed with 100ml solution of UT-P 0.02% once a day for a maximum of 5 instillations.

SUMMARY:
It is the first clinical study aimed at assessing the safety and tolerability of UT-P as routine rinsing and bacterial decolonization solution device for urinary catheters. The study will be conducted in hospitalized adult patients who had an urethral or suprapubic catheter in place for longer than two consecutive weeks and who are able to provide written consent.

This is an open-label prospective observational cohort study. No comparative control group is planned as no other preventing infection solution is commercially available at this time.

DETAILED DESCRIPTION:
The objective of this study is to assess the tolerability and safety of Uro-Tainer® Polihexadine 0.02% intended as routine rinsing and bacterial decolonization of urinary catheters in long-term catheterized patients. After each instillation patients will be assessed for vital signs, skin reactions and other symptoms suggesting intolerance or sensitivity and/or allergic reaction. In addition, pain will be assessed in the first 5 patients and any other patients with sustained pain sensation in the bladder.

Catheters will be rinsed by gravity feed with 100ml solution of UT-P 0.02% once a day for a maximum of 5 instillations. A minimum interval of 24 hours must be guaranteed for the enrolment of the first 5 patients and their first irrigation with the investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a sustained pain sensation in the bladder (for the first five patients).
* Patients staying as inpatients with long-term (> 2 weeks) urethral or suprapubic catheters.

  * Age > 18 years
  * Ability to read, write and speak German or French
  * Women of child bearing potential must test negative on standard urine pregnancy test two weeks prior to the start of the study and must agree to practice appropriate contraceptive methods until the end of the study (e.g. oral contraceptive, IUD, intra-muscular contraceptive, abstinence).
  * Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent approved by the cantonal Ethics Committee (IEC) prior to all evaluations

Exclusion Criteria:

* Symptomatic UTI
* Hematuria
* Fever (tympanic temperature > 38.5°C)
* Surgical intervention to genito-urinary tract in the last 6 months
* Patients receiving any other concurrent catheter irrigation
* Known allergy or sensitivity to any of the ingredients in Uro-Tainer® Polihexanide 0.02%
* Known allergy or sensitivity to chlorhexidine
* Pregnancy or Lactation
* Simultaneous participation in another interventional trial
* Administration of any other catheter irrigation 1 week prior to study
* Administration of any of the following medications 4 weeks prior to study entry, unless they have been used at a stable regimen : antibiotics, antipyretics, antihistamines, medications susceptible to cause an autonomic response or to mask an allergic reaction.
* For the first five patients: impaired pain sensation in the bladder for the first five patients: Administration of any antipyretics and analgesic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
to assess the tolerability of Uro-Tainer® Polihexanide 0.02% | Day 1, Day 2, Day 3, Day 4, Day 5
  Change in Visual Analogue Scale (VAS) Score for patients with sustained pain sensation in the bladder Bladder spasms Blood pressure (change in SBP ≥ 40 mmHg is a discontinuation criterion, see 7.4.3) Heart rate Change in tympanic temperature Urine Dipstick (LEU) Occurrence of Flushing Occurrence of Sweating

SECONDARY OUTCOMES:
To assess the safety of Uro-Tainer® Polihexanide 0.02% in long-term catheterized patients | Day 1, Day 2, Day 3, Day 4, Day 5
  Adverse Events
  * Urticaria
  * Exanthema
  * Any other signs and symptoms associated with allergic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Pannek, Prof., Principal Investigator — Schweizer Paraplegikerzentrum Nottwil
Locations (5):
- Universitair Ziekenhuis, Ghent, Belgium
- Kliniken-Beelitz GmbH, Beelitz-Heilstätten, Germany
- Switzerland (3):
  - Schweizerisches Paraplegikerzentrum, Basel, Canton of Basel-City
  - Schweizer Paraplegikerzentrum, Nottwil, Canton of Lucerne
  - Rehaklinik, Valens, Canton of St. Gallen

REFERENCES:
- [Derived] Pannek J, Everaert K, Mohr S, Vance W, Van der Aa F, Kesselring J. Tolerability and safety of urotainer(R) polihexanide 0.02% in catheterized patients: a prospective cohort study. BMC Urol. 2020 Jul 8;20(1):92. doi: 10.1186/s12894-020-00650-1. PMID 32641131